CLINICAL TRIAL: NCT00599365
Title: Impact of a Pharmacist's Collaborative Management, Adherence,and Medication Education Program (CAMP) in an Ambulatory Renal Clinic
Brief Title: Impact of CAMP in an Ambulatory Renal Clinic
Acronym: CAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Nelson Chee Pharm.D, VA Medical Center, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H45161-31657-01; T0986
Record Dates: First submitted 2008-01-04; First posted 2008-01-23 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Kidney Disease
Keywords: adherence; pharmacist intervention; persistence; renal clinic; pill count
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacy Care arm (Experimental): The pharmacist:
  * will take all the patient's medication bottles, and give medication boxes filled with medications in the order the patient should take them in.
  * will need to obtain a complete list of medications.
  * will teach the patient about the medications.
  * will provide a medication schedule, and other papers about the medications.
  * will count the pills in the medication boxes.
  * will review all the medications with the patient and answer any question.
  * will check to see if the medication is working for the patient.
  * will work with the patient's kidney doctor to adjust medications if needed.
  * will give the medication boxes filled with medications to take home.
  Interventions: Other: Pharmacy care arm
- Control (No Intervention): The pharmacist:
  * will obtain a complete list of medications.
  * will count the pills in the patients' medication bottles.
  * will inform patients to take their medications from these bottles.

INTERVENTIONS:
Other: Pharmacy care arm — * The pharmacist will take all your medication bottles, and give you medication boxes filled with your medications in the order you should take them in.
  * You will need to give a complete list of medications to the pharmacist.
  * You will need to describe how you take these medications.
  * The pharmacist will teach you about the medications. This includes side effects, drug interactions, and directions.
  * The pharmacist will give you a medication schedule, and other papers about your medications.
  Arms: Pharmacy Care arm

SUMMARY:
The purpose of this study is to see if a pharmacist can help patients understand how he/she should be taking their medications. The study is also being done to see if meeting with the pharmacist can help patients better control chronic kidney disease and the medical problems that can occur.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a serious condition associated with premature mortality, decrease quality of life, and increase health-care costs. An estimated 19 million Americans (1 in 9 US adults) have non-dialysis dependent CKD (Stages 1-4).1 The health care expenditures for caring for patients with CKD are substantial. According to Centers for Medicare and Medicaid Services (CMS), the estimated annual health cost per patient for managing patients with CKD is markedly higher ($28,000) compared to the costs for caring for diabetic patients ($10,000 per patient) and heart failure patients ($5000 per patient). 2 According to the National Kidney Foundation, as renal function declines, the number of renal complications, notably high blood pressure, anemia, malnutrition, and mineral and bone disorders, increases along with the severity. A large proportion of patients with CKD also develop multiple co-morbidities, particularly hypertension, diabetes, and hyperlipidemia. Fortunately, accumulating evidence indicates that treatment of earlier stages of chronic kidney disease can prevent the development of kidney failure (Stage 5)3. In addition, early prevention of cardiovascular risk factors in patients with CKD may reduce cardiovascular events before and after the onset of kidney failure.3 Because many patients, particularly in the later stages of CKD, have multiple renal complications and chronic co-morbidities, these patients are potentially at high risk of medication non-adherence and non-persistence (defined as premature discontinuation of medication therapy). Studies have demonstrated that patients with chronic diseases typically take only 50% of prescribed doses of medication, leading to increased disease severity, clinic visits, and hospital admissions, resulting in substantial healthcare expenditures.4,5 In the United States alone, the cost of illness, due to non-adherence was estimated to be $170 billion per year.6 In addition, the associated total cost of treating the complications resulting from poor adherence in dialysis and transplant patients exceeds $950 million.7 Potential barriers to medication adherence for patients with chronic diseases include, but are not limited to, complex medication regimens, multiple drug doses, treatment of asymptomatic conditions, and cognitive factors. Although not well-studied in pre-dialysis patients, limited data suggests that important causes of medication non-adherence in chronic dialysis patients include inadequate prescription coverage or high medication costs, lack of transportation, and adverse effects. 8

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for enrollment if they are > 18 year old men or women receiving care from the VAMCSF Renal Clinic with a documented diagnosis of CKD stage 2-5, and are receiving pharmacological treatment for one or more medical conditions of CKD, including hypertension, diabetes, CKD-mineral and bone disorders, and/or anemia of chronic disease.

Exclusion Criteria:

Patients will be excluded from the study if they obtain medications prescribed for the above medical conditions from a facility outside the VAMCSF, are enrolled in Medi-Set clinic, are kidney transplant patients, are diagnosed with CKD stage 1, require assistance in the administration of their medications (i.e. caregiver), lack adequate transportation to clinic, and/or lack telephone access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
MPR cumulative persistence rates pill counts blood glucose HgbA1c hemoglobin concentration iron ferritin transferrin saturation SBP/DBP corrected calcium phosphorous calcium-phosphorus product uAlb/Cr eGFR. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Chee, Pharm.D, Principal Investigator — VA Medical Center San Francisco
Locations (1):
- VA Medical Center San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Chen RA, Scott S, Mattern WD, Mohini R, Nissenson AR. The case for disease management in chronic kidney disease. Dis Manag. 2006 Apr;9(2):86-92. doi: 10.1089/dis.2006.9.86. PMID 16620194
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Haynes RB, Yao X, Degani A, Kripalani S, Garg A, McDonald HP. Interventions to enhance medication adherence. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD000011. doi: 10.1002/14651858.CD000011.pub2. PMID 16235271
- [Background] Kripalani S, Yao X, Haynes RB. Interventions to enhance medication adherence in chronic medical conditions: a systematic review. Arch Intern Med. 2007 Mar 26;167(6):540-50. doi: 10.1001/archinte.167.6.540. PMID 17389285
- [Background] Dezii CM. Medication noncompliance: what is the problem? Manag Care. 2000 Sep;9(9 Suppl):7-12. No abstract available. PMID 11729418
- [Background] Loghman-Adham M. Medication noncompliance in patients with chronic disease: issues in dialysis and renal transplantation. Am J Manag Care. 2003 Feb;9(2):155-71. PMID 12597603
- [Background] Reddy SS, Holley JL. Management of the pregnant chronic dialysis patient. Adv Chronic Kidney Dis. 2007 Apr;14(2):146-55. doi: 10.1053/j.ackd.2007.01.005. PMID 17395117
- [Background] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639
- [Background] Murray MD, Young J, Hoke S, Tu W, Weiner M, Morrow D, Stroupe KT, Wu J, Clark D, Smith F, Gradus-Pizlo I, Weinberger M, Brater DC. Pharmacist intervention to improve medication adherence in heart failure: a randomized trial. Ann Intern Med. 2007 May 15;146(10):714-25. doi: 10.7326/0003-4819-146-10-200705150-00005. PMID 17502632
- [Background] Chisholm MA, Mulloy LL, Jagadeesan M, Martin BC, DiPiro JT. Effect of clinical pharmacy services on the blood pressure of African-American renal transplant patients. Ethn Dis. 2002 Summer;12(3):392-7. PMID 12148711
- [Background] Allenet B, Chen C, Romanet T, Vialtel P, Calop J. Assessing a pharmacist-run anaemia educational programme for patients with chronic renal insufficiency. Pharm World Sci. 2007 Feb;29(1):7-11. doi: 10.1007/s11096-005-4800-4. PMID 17268940
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Rodbard HW, Blonde L, Braithwaite SS, Brett EM, Cobin RH, Handelsman Y, Hellman R, Jellinger PS, Jovanovic LG, Levy P, Mechanick JI, Zangeneh F; AACE Diabetes Mellitus Clinical Practice Guidelines Task Force. American Association of Clinical Endocrinologists medical guidelines for clinical practice for the management of diabetes mellitus. Endocr Pract. 2007 May-Jun;13 Suppl 1:1-68. doi: 10.4158/EP.13.S1.1. No abstract available. PMID 17613449
- [Background] Halpern MT, Khan ZM, Schmier JK, Burnier M, Caro JJ, Cramer J, Daley WL, Gurwitz J, Hollenberg NK. Recommendations for evaluating compliance and persistence with hypertension therapy using retrospective data. Hypertension. 2006 Jun;47(6):1039-48. doi: 10.1161/01.HYP.0000222373.59104.3d. Epub 2006 May 1. No abstract available. PMID 16651464
- [Background] Sikka R, Xia F, Aubert RE. Estimating medication persistency using administrative claims data. Am J Manag Care. 2005 Jul;11(7):449-57. PMID 16044982
- [Background] American Diabetes Association. Standards of medical care in diabetes--2007. Diabetes Care. 2007 Jan;30 Suppl 1:S4-S41. doi: 10.2337/dc07-S004. No abstract available. PMID 17192377